CLINICAL TRIAL: NCT01388439
Title: Pharmacokinetics of Oseltamivir in Newborns and Infants
Status: Completed | Type: Observational
Sponsor: St. Louis Children's Hospital (Other)
Collaborators: Genentech, Inc. (Industry); Washington University School of Medicine (Other)
Responsible Party: Christopher McPherson, St. Louis Children's Hospital
Other Study IDs: TAM 027
Record Dates: First submitted 2011-06-24; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-06

CONDITIONS: Prematurity of Fetus
Keywords: oseltamivir; influenza; neonate; premature; pharmacokinetics
MeSH Terms: conditions — Influenza, Human; Premature Birth | interventions — Oseltamivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two whole blood samples (0.5 mL) were obtained at steady state (day 3 of therapy or later), collected in K3EDTA mini-collection tubes labeled with a sample identification number. Plasma specimens were separated by centrifugation of 1500 g for 10 minutes at 4 degrees Celsius within 60 minutes of sample collection. Plasma supernatant was transferred into a cryovial labeled with the same sample identification number. Cryovials were immediately stored at -70 degrees Celsius. Sample obtainment and processing was directly supervised by the principle investigator.
  The blood samples are currently being stored at -70 degrees Celsius in a research laboratory operated by medical faculty of the Washington University School of Medicine Department of Pediatrics Division of Infectious Diseases in the McDonnell Medical Sciences Building.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oseltamivir exposure: One infant in the Neonatal Intensive Care Unit (NICU) at St. Louis Children's Hospital experienced respiratory decompensation and tested positive for influenza virus type A by fluorescent antibody stain performed on a nasopharyngeal swab. This infant received treatment doses of oseltamivir. Subsequently, 27 other infants received oseltamivir prophylaxis for exposure to influenza virus type A. Exposed infants were those who shared a primary medical team, nursing care, respiratory therapist, physical therapist, or occupational therapist with the influenza A positive infant. Prophylaxis was deemed necessary by the attending neonatologist after consultation with the Infectious Diseases Division of the Department of Pediatrics at the Washington University School of Medicine.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Treatment dose was oseltamivir 3 mg/kg/dose by mouth (PO) twice daily. Prophylactic dose was oseltamivir 1 mg/kg/dose PO once daily to infants < 28 weeks postmenstrual age (PMA), 1 mg/kg/dose PO twice daily to infants 28 - 38 weeks PMA, and 3 mg/kg/dose PO once daily to infants > 38 weeks PMA. Dosing in infants < 28 weeks PMA was chosen based on unpublished data from Acosta et al. This data was obtained from phone contact with Dr. Peter Gal, co-author of the study. Dosing in infants 28 - 38 weeks PMA was chosen based on published data from Acosta et al.1 Dosing in infants > 38 weeks PMA and less than 3 months postnatal age was chosen based on data from Kimberlin et al. Dosing in infants > 38 weeks PMA and greater than 3 months postnatal age was per the recommendations of the Advisory Committee on Immunization Practices of the United States Department of Health and Human Services.

SUMMARY:
Oseltamivir dosing in infants < 3 months of age is based on a single pharmacokinetic study in 20 infants from a single center. This dataset is limited by a lack of robustness, because only 1 sample was collected from each participant. The investigators obtained two blood samples each from infants receiving oseltamivir after obtaining informed consent from the infant's parents. The investigators propose to analyze the blood samples to determine the amount of oseltamivir in the infant's blood. Measurement of these values will increase the understanding of the absorption and elimination of oseltamivir in preterm and term infants, and improve our ability to provide the correct doses to this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* All neonates and infants in the NICU at St. Louis Children's Hospital who received oseltamivir for treatment of or exposure to influenza virus type A were considered eligible for this study.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: One infant in the Neonatal Intensive Care Unit (NICU) at St. Louis Children's Hospital experienced respiratory decompensation and tested positive for influenza virus type A by fluorsescent antibody stain performed on a nasopharyngeal swab. This infant received treatment doses of oseltamivir. Subsequently, 27 other infants received oseltamivir prophylaxis for exposure to influenza virus type A. Exposed infants were those who shared a primary medical team, nursing care, respiratory therapist, physical therapist, or occupational therapist with the influenza A positive infant. Prophylaxis was deemed necessary by the attending neonatologist after consultation with the Infectious Diseases Division of the Department of Pediatrics at the Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Oseltamivir pharmacokinetics in neonates and infants | Two sample points, one 0-3 hours (baseline) and one 3-24 hours post dose
  Pharmacokinetic parameters calculated for individual subjects will include apparent distribution volume and elimination half-life of oseltamivir (OST) and OST carboxylate (CBX). Area under the plasma concentration versus time curve (AUC) of OST and OST CBX will be determined using the trapezoidal method. A population pharmacokinetic model will be generated based on pooled pharmacokinetic data (2-compartment model for OST and 1-compartment model for OST CBX) utilizing maximum likelihood estimation. A weight-based dosing table will be generated to provide AUC exposures comparable to adults.

SECONDARY OUTCOMES:
Oseltamivir target level attainment | Two sample points, one 0-3 hours (baseline) and one 3-24 hours post dose
  OST target level attainment of the currently recommended dosing regimen in neonates and infants will be calculated. Currently recommended doses were utilized for all neonates and infants in our cohort. The target level attainment in this cohort will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Louis Children's Hosptial, St Louis, Missouri, United States

REFERENCES:
- [Background] Acosta EP, Jester P, Gal P, Wimmer J, Wade J, Whitley RJ, Kimberlin DW; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Oseltamivir dosing for influenza infection in premature neonates. J Infect Dis. 2010 Aug 15;202(4):563-6. doi: 10.1086/654930. PMID 20594104
- [Background] Fiore AE, Fry A, Shay D, Gubareva L, Bresee JS, Uyeki TM; Centers for Disease Control and Prevention (CDC). Antiviral agents for the treatment and chemoprophylaxis of influenza --- recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2011 Jan 21;60(1):1-24. PMID 21248682